CLINICAL TRIAL: NCT00509353
Title: Irinotecan and Vincristine With 131I-MIBG Therapy for Resistant/Relapsed High-Risk Neuroblastoma, A Phase I Study
Brief Title: N2004-06: Irinotecan and Vincristine With 131I-MIBG Therapy for Resistant/Relapsed High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Araz Marachelian, Medical Director, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558042; P01CA081403 (NIH); N2004-06 (Other: NANT Consortium); NANT-Draximage-2007-01 (Other: Draximage)
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Irinotecan; Vincristine; 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: irinotecan hydrochloride; Drug: vincristine sulfate; Radiation: iobenguane I 131

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: vincristine sulfate
Radiation: iobenguane I 131

SUMMARY:
RATIONALE: Radioactive drugs, such as iodine I 131 metaiodobenzylguanidine (MIGB), may carry radiation directly to tumor cells and not harm normal cells. Drugs used in chemotherapy, such as irinotecan and vincristine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving iodine I 131 MIGB together with irinotecan and vincristine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of iodine I 131 MIGB when given together with irinotecan and vincristine in treating young patients with resistant or relapsed high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of iodine I 131 metaiodobenzylguanidine when given in combination with fixed-dose irinotecan hydrochloride and vincristine in young patients with refractory or relapsed high-risk neuroblastoma.
* To determine the dose-limiting toxicities of iodine I 131 metaiodobenzylguanidine when combined with fixed-dose irinotecan hydrochloride and vincristine.

Secondary

* To determine if there is a therapeutic response to this regimen.

OUTLINE: This is a multicenter, dose-escalation study of iodine I 131 metaiodobenzylguanidine (^131I-MIBG).

Patients receive ^131I-MIBG IV over 1½-2 hours on day 1, vincristine IV on days 0 and 7, and irinotecan hydrochloride IV over 1 hour on days 0-4 and 7-11. Treatment repeats every 56 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Must have a diagnosis of neuroblastoma by histologic verification and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines
* Must have high-risk neuroblastoma AND meets at least one of the following criteria:

  * Recurrent or progressive disease at any time

    * Biopsy not required, even if there is partial response to intervening therapy
  * Refractory disease (i.e., less than a partial response to frontline therapy, including a minimum of 4 courses of chemotherapy)

    * Biopsy not required
    * If the patient has not had previous myeloablative therapy, preference will be given to NANT-2001-02 (iodine I 131 metaiodobenzylguanidine [^131I-MIBG] + CEM)
  * Persistent disease after at least a partial response to frontline therapy (i.e., patient still has residual disease by MIBG scan, CT/MRI scan, or bone marrow)

    * Biopsy required (bone marrow biopsy included) of at least one residual site demonstrating viable neuroblastoma
    * If the patient has not had previous myeloablative therapy, preference will be given to NANT-2001-02 (^131I-MIBG + CEM)
* Must have evidence of MIBG uptake into tumor at ≥ 1 site within 4 weeks prior to study entry and subsequent to any intervening therapy
* Must have autologous hematopoietic stem cell product available and it must be free of tumor cell contamination (0 tumor cells /1,000,000 nucleated cells), cryopreserved, and available for re-infusion after ^131I-MIBG treatment, if immunocytology has been performed on the stem cell product

  * If immunocytology has not been performed on the stem cell product, then bilateral bone marrow aspirates and biopsies must have been negative by morphology within 4 weeks before or after the stem cell collection
  * If the patient had no bone marrow disease documented at diagnosis or at any time prior to peripheral blood stem cell (PBSC) harvest then the criteria for bilateral bone marrow aspirates/biopsies is waived
  * The minimum dose is as follows:

    * Purged PBSC 2.0 x 10^6 viable CD34+ cells/kg

      * Immuno-magnetically purged cells are permitted
    * Unpurged PBSC 2 x 10^6 CD34+ cells/kg (minimum is same for PBSC from identical twin)
  * Cells from identical twins are permitted

    * Other allogeneic cells are not allowed
  * CD34+ selected cells are not permitted

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Lansky or Karnofsky performance status ≥ 50%
* Life expectancy ≥ 6 weeks
* Hemoglobin ≥ 8 g/dL (transfusion allowed)
* ANC ≥ 750/μL (no hematopoietic growth factors within 7 days of starting irinotecan hydrochloride)
* Platelet count ≥ 50,000/μL (transfusion independent, defined as no platelet transfusion for 2 weeks)
* Glomerular filtration rate (GFR) or creatinine clearance ≥ 60 mL/min OR age-adjusted serum creatinine ≤ 1.5 x normal, according to the following:

  * 0.8 mg/dL (≤ 5 years of age)
  * 1.0 mg/dL (6 to 10 years of age)
  * 1.2 mg/dL (11 to 15 years of age)
  * 1.5 mg/dL (≥ 16 years of age)
* Total bilirubin ≤ 1.5 x normal for age
* ALT and AST < 3 x normal for age
* All post-menarchal females must have a negative beta-HCG
* Males and females of reproductive age and childbearing potential must use effective contraception for the duration of study participation
* Ejection fraction ≥ 55% by echocardiogram or radionuclide MUGA OR fractional shortening ≥ 27% by echocardiogram
* Normal lung function
* Patients with other ongoing serious medical issues must be approved by the study chair prior to study registration

Exclusion criteria:

* Pregnancy or breast feeding
* Dyspnea at rest, exercise intolerance, pleural effusion, or oxygen requirement
* Disease of any major organ system that would compromise the patient's ability to withstand therapy
* Documented allergy to third generation cephalosporins
* Active diarrhea (defined as ≥ grade 2 per CTCAE v3)
* Active or uncontrolled infection, including C. difficile

  * Patients on prolonged antifungal therapy are eligible if suspected radiographic lesions are culture and biopsy negative and patient meets other organ function criteria
* Patients and/or families who are physically and psychologically unable to cooperate with the radiation safety isolation
* Patient weight that would require exceeding a maximum total allowable dose of ^131I-MIBG (per institutional guidelines)
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy before study entry
* At least 3 weeks since prior myelosuppressive or biologic therapy
* At least 2 weeks since prior radiation therapy

  * Radiation therapy should not be given to the only site of measurable or evaluable disease
* At least 3 months since prior large field radiation therapy (i.e., craniospinal radiation therapy, total lung radiation therapy, or radiation therapy to > 50% of marrow space)
* At least 3 months since prior autologous stem cell transplantation

  * Must meet adequate bone marrow function postmyeloablative therapy
* At least 7 days since prior cytokines or hematopoietic growth factors
* Prior irinotecan hydrochloride and vincristine therapy allowed provided the patient recovered to adequate bone marrow function as specified in the protocol

Exclusion criteria:

* Prior ^131I-MIBG
* Prior external beam radiation therapy to the liver or kidneys
* Prior allogeneic stem cell transplantation
* Prior whole abdominal radiation therapy, total-body irradiation, or local radiation therapy that includes any of the following:

  * 1,200 cGy to more than 33% of both kidneys (patient must have at least one kidney that has not exceeded the dose/volume of radiation listed)
  * 1,800 cGy to more than 30% of liver and/or 900 cGy to more than 50% of liver
* Other concurrent cancer chemotherapy or immunomodulating agents (including steroids)

  * Steroids may be used in the prevention and treatment of transfusion/infusion reactions and for the treatment of edema associated with CNS lesions
* Concurrent palliative radiotherapy to localized painful lesions
* Concurrent aprepitant (Emend)
* Concurrent ketoconazole or St. John's wort
* Medications that interfere with MIBG uptake during the week prior to or after MIBG therapy
* Concurrent enzyme-inducing anticonvulsants (e.g., phenobarbital, phenytoin, or carbamazepine)

  * Nonenzyme-inducing anticonvulsants (e.g., Keppra) may be allowed
* Concurrent hemodialysis
* Any other concurrent anticancer agents or radiation therapy

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of 131I-MIBG given in combination with fixed-dose irinotecan/vincristine to children with high-risk refractory/relapsed neuroblastoma. | Tolerability will be assessed throughout the study.
To determine the dose limiting toxicities of 131I-MIBG combined with irinotecan/vincristine. | Adverse events, clinically significant changes in laboratory results, and vital signs, to be measured throughout the study.

SECONDARY OUTCOMES:
Within the confines of a Phase I study, to determine if there is a therapeutic response to this regimen. | Disease response will be evaluated at baseline, prior to each cycle and at the end of treatment.
  Disease response will be evaluated by any of the following CT, MRI, MIBG, Bone Marrow, Urine Catecholamines at baseline, prior to each cycle and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, Principal Investigator — UCSF Medical Center at Parnassus
Locations (12):
- United States (12):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin